CLINICAL TRIAL: NCT02258672
Title: Effects of a Preoperative Rehabilitation Program on the Recovery of Patients Undergoing Surgery for Lumbar Spinal Stenosis: a Feasibility Study.
Brief Title: Preoperative Rehabilitation for Patients Undergoing Surgery for Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Fonds de soutien au démarrage de projets en collaboration (CSSSTR) (Unknown); Fonds pour la Recherche Clinique de l'UQTR (Unknown)
Responsible Party: Principal Investigator, Martin Descarreaux, DC, PhD, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UQTR-CSSSTR 2014
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Preoperative rehabilitation; Minimally invasive surgery; Functional capacity
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation program (Experimental): Participants will be physically trained before undergoing surgery
  Interventions: Other: Prehabilitation program
- Control (No Intervention): Patients will follow the normal course of care provided by the hospital

INTERVENTIONS:
Other: Prehabilitation program — Progressive and individualized physical training aimed at improving core muscles strength and endurance as well as spinal stability.
  Arms: Prehabilitation program

SUMMARY:
The purpose of the present study is to evaluate the effectiveness of a prehabilitation program on the recovery of patients undergoing a minimally invasive surgery for degenerative lumbar spinal stenosis. To do so, 40 participants will be recruited and randomized into two groups; intervention or control group. Participants in the intervention group will take part in a physical training program, three times a week for six weeks before undergoing surgery. The exercise program will be supervised and will aim at improving core muscles strength and endurance as well as spine stability. It is hypothesized that the prehabilitation program will significantly improve disability and pain intensity reported by patients after surgery. Ultimately, this study aims to improve health care of patients awaiting lumbar surgery but its results may also impact the management of patients awaiting spine surgery for various conditions.

ELIGIBILITY:
Inclusion Criteria:

To be affected by degenerative lumbar spinal stenosis and to be awaiting minimally invasive surgery for the lumbar spinal stenosis

Exclusion Criteria:

Non-degenerative spinal stenosis, arthritic conditions (except for facet arthrosis), impaired cognitive function, spinal instability and disagreement from the treating neurosurgeon for the patient to take part in the preadaptation programme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in disability | baseline, week 6, week 10, week 18, week 30
  Oswestry Disability Index

SECONDARY OUTCOMES:
Change from Baseline in pain intensity | baseline, week 6, week 10, week 18, week 30
  Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC, PhD, Study Director — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

REFERENCES:
- [Derived] Marchand AA, Suitner M, O'Shaughnessy J, Chatillon CE, Cantin V, Descarreaux M. Effects of a prehabilitation program on patients' recovery following spinal stenosis surgery: study protocol for a randomized controlled trial. Trials. 2015 Oct 27;16:483. doi: 10.1186/s13063-015-1009-2. PMID 26507388